CLINICAL TRIAL: NCT05974956
Title: Effect of a Nursing Teaching Protocol on Mastitis Prognosis: Quasi-Experimental Research Design
Acronym: Mastitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amna A. Desouky, MD, Assistant professor of Medical Surgical Nursing, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Mastitis prognosis
Record Dates: First submitted 2023-07-02; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Mastitis
MeSH Terms: conditions — Mastitis

STUDY DESIGN:
Intervention Model Description: Quasi experimental research design that test for change through manipulation of the independent variable. However, in this study, it lacks one of the three key properties of an experimental design "randomization".
  The dependent variables (mastitis knowledge, self -care practice, pain level, and complications associated with mastitis) were measured and compared at base line for both control and study groups, then intervention was introduced to the study group. After three weeks; the dependent variables for both groups were evaluated to test the difference.
Who Masked: Outcomes Assessor
Masking Description: Medical researcher "N" assessed the prognosis of mastitis using tool IV" mastitis prognosis sheet for all patients "control - study" at follow up without knowing the study group who received the nursing teaching protocol
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group exposed to routine care.
- Study group (Experimental): The study group received the sessions of "mastitis care teaching protocol".
  Interventions: Other: Mastitis care teaching protocol

INTERVENTIONS:
Other: Mastitis care teaching protocol — It was developed by the authors based on previous similar studies, articles and library resources. It was introduced to the study group in the form of face to face sessions plus a hand out copy. It consisted of three parts; (1): Theoretical part about mastitis (definition, types, clinical manifestation, possible causes, diagnosis and management). (2):Self-care practices, and (3):Recommendations regarding dietary measures, rest, medication and follow up.
  Arms: Study group

SUMMARY:
Aim: Evaluate the effect of a nursing teaching protocol on mastitis prognosis. Research design: Quasi-experimental research design was utilized. A convenient sample of sixty adult female patients diagnosed with mastitis, Patients divided equally into two groups(study and control) thirty for each.

DETAILED DESCRIPTION:
The study was conducted in the breast unit in general surgery department at Main Assiut University Hospital. A convenient sample of sixty adult female patients diagnosed with mastitis, their ages range from 20 to 65years old. Patients divided equally into two groups; thirty for each. Both groups had been assessed at base line using the following tools:

Tool (I): An interview questionnaire sheet Tool (II):Mastitis self-care practices Tool (III): Numeric pain rating scale Tool (IV): Mastitis prognosis sheet

The control group exposed to routine care and study group received mastitis teaching protocol. After three weeks; both groups had been reassessed by the same tools.

Data analysis had been performed by using the Statistical Package for the Social Sciences (SPSS) Categorical variables described by number and percent (N, %). Continuous variables described by mean and standard deviation (Mean, SD). Chi-square test and Fisher exact test used to compare between categorical variables .T-test and Pearson's chi-square used to appear the association between patients' knowledge, practice, and mastitis prognosis before implementation of nursing teaching protocol and three weeks post.

ELIGIBILITY:
Exclusion Criteria:

1. Mental health problems
2. Visual or hearing problems
3. Uncooperative

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Inclusion criteria:
  1. Adult women
  2. Age from 20 to 65 yrs.
  3. Clinical diagnosis of mastitis
  4. Lactational or non-lactational mastitis
Enrollment: 60 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Compare the difference between the mean knowledge of participants (study and control groups) regarding mastitis care and management at base line & follow up after three weeks. | Base line assessment: Is the first assessment --------- Follow up assessment:: after three weeks
  The knowledge of participants(study and control groups) regarding mastitis care and management had been assessed twice( base line - follow up) using: Tool I: An interview questionnaire sheet (part 2)
  Tool I: It was structured by authors and reviewed by a panel of experts in General Surgery and Medical -Surgical Nursing.
  Each answered question scored from 0 to 3 marks as follows; 3 marks for complete correct answer, 2 marks for incomplete correct answer, 1 mark for incorrect answer and zero for not known answer.
  The range of total score lies between 0-30, the scoring system interpreted in the results into satisfactory and unsatisfactory; satisfactory: if the total knowledge score is ≥ 60% and unsatisfactory if the total knowledge score is < 60%.
Compare the difference between the mean practice of participants (study and control groups) regarding mastitis care and management at base line & follow up after three weeks. | Base line assessment: Is the first assessment --------- Follow up assessment:: after three weeks
  The performance of participants (study and control groups) regarding mastitis care and management had been assessed twice (baseline- follow up) using: Tool II: "Mastitis self-care practices".
  Tool II: It was structured by authors and reviewed by a panel of experts in General Surgery and Medical -Surgical Nursing.
  Scoring:
  A total score of 60% or higher considered as adequate self-care practices and less than 60% considered as inadequate. Three points scale used to grade the steps. Two points for doing correctly. One point for doing incorrectly and zero point for not doing at all.

SECONDARY OUTCOMES:
Pain level using Numeric Pain Rating scale | Base line assessment: Is the first assessment --------- Follow up assessment:: after three weeks
  Pain level as a symptom of mastitis was measured at base line using Tool III: Numeric Pain rating scale for both study and control groups.
  It was asked from each patient to rate pain level from 0 to10 with understanding that 0 is equal to no pain and 10 is equal to worst possible pain.
  At follow up "third week" pain level was measured again for both study and control groups with the same scale to test for change.
Number of participants(study -control) who discontinued breast feeding | At the third week from base line assessment.
  Lactating women in either groups (study -control) reported that they discontinued nursing their babies.
  This outcome was evaluated by using tool IV: "Mastitis prognosis sheet" that had been structured by authors and reviewed by a panel of experts in General Surgery and Medical -Surgical Nursing.
Number of participants (study -control) who completely cured from mastitis | At the third week from base line assessment.
  Inflamed breast was evaluated for both groups (study- control), If it resolved and returned to normal condition or not.
  This outcome was evaluated clinically (signs & symptoms) by using tool IV: "Mastitis prognosis sheet" that had been structured by authors and reviewed by a panel of experts in General Surgery and Medical -Surgical Nursing.
Number of participants (study -control) who their condition complicated with formation of breast abscess. | At the third week from base line assessment.
  Breast abscess is a complication of mastitis that will be formed within the inflamed breast tissue.
  This outcome was evaluated clinically (signs and symptoms) by using tool IV: "Mastitis prognosis sheet" that had been structured by authors and reviewed by a panel of experts in General Surgery and Medical -Surgical Nursing.
Number of mastitis recurrence among participants(study -control) . | At the third week from base line assessment.
  The inflamed breast tissue re-inflamed again for the second time.
  This outcome was evaluated clinically (signs and symptoms) by using tool IV: "Mastitis prognosis sheet" that had been structured by authors and reviewed by a panel of experts in General Surgery and Medical -Surgical Nursing.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Yes: There is a plan to make IPD and related data dictionaries available.
Supporting Information: SAP, CSR